CLINICAL TRIAL: NCT06012825
Title: Pediatric Physical Activity (PePA): Understanding Best Practices in Implementing Physical Activity for Patients Diagnosed With Childhood Cancer
Brief Title: Pediatric Physical Activity for Children With Cancer
Acronym: PePA
Status: Completed | Type: Observational
Sponsor: University of Hawaii (Other)
Collaborators: Hawaii Pacific Health (Other); University of Hawaii Cancer Research Center (Other)
Responsible Party: Principal Investigator, Paulette M. Yamada, Associate Professor, University of Hawaii
Other Study IDs: 2021-084
Record Dates: First submitted 2023-05-04; First posted 2023-08-28 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pediatric Cancer; Physical Activity
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physical Activity (PA) Round 1: All enrollees will have the opportunity to attend virtual PA sessions.
  Interventions: Behavioral: Physical Activity
- Physical Activity Round 2: This second cohort is the 2nd round of intervention, which allows participants to enroll for another round, and/or newly recruited patients will have the opportunity to participate.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — The program will consist of 2 consecutive rounds of 12-week programming, 2x/week for 60 minutes on a Health Insurance Portability and Accountability Act (HIPAA)-compliant Zoom account. The PA program will be structured to ensure equivalent "PA doses" are provided. This will be done by allocating time to a warm-up (5 min), an introduction and demonstration of the activity (5 min), the PA (30 min), cool down and stretching (5 min). Time will also be devoted for interaction to develop rapport, transition to the next activity, and to handle internet connectivity issues (15 min).

SUMMARY:
The goal of this pilot study is to test the feasibility and participant adherence (pediatric patients diagnosed with childhood cancer) to a virtual, 12-week physical activity program.

The aims of this project are to:

1. Determine the feasibility of administering the program and patient acceptability.
2. Report program adherence and completion rates.
3. Explore trends on the impact of a virtual PA intervention on psychosocial health and physical fitness.

Participants will undergo pre- and post-assessments including measurements of fitness, self-reported fatigue and depression symptoms, social support, and current amount of physical activity. Patients will then be invited to participate in two consecutive, 12-week virtual physical activity interventions with similar-aged peers (2x/week, 60 minutes/session) over 2 rounds.

DETAILED DESCRIPTION:
It is critical for childhood cancer patients to maintain a physical activity (PA) regime as they are at an increased risk of developing co-morbidities. PA engagement is associated with positive psychosocial outcomes, and it has the potential to improve cardiopulmonary and musculoskeletal function. Patients will be enrolled and will undergo baseline assessments of fitness and quality of life as part of their standard care, and additional measures that include fatigue, depression, social support, and PA volume will be measured. Patients will be invited to participate in a 12-week virtual PA intervention with similar-aged peers (2x/week, 60 minutes/session). Patients will be led through activities that are culturally relevant and age-appropriate. At the end of the 12-week intervention, the same tests will be completed. The patients will have an opportunity to receive 2 interventions. A mixed method design will be used, where quantitative data will include information related to feasibility, PA volume, physical fitness, and psychosocial health measures, and qualitative data will be collected from the patients during the focus groups.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with cancer
* Ability to connect to virtual sessions 2x/week
* English literacy
* Having guardian consent and patient assent.
* Eligible patients will be those who do not require physical therapy (i.e., able to dress, ambulate) and will be physically able to participate, as determined by therapy staff.

Exclusion Criteria:

* Not having been diagnosed with cancer.
* Inability to communicate in English
* Requires physical or occupational therapy.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients referred by their physician at a primary care facility.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Enrollment | Tracked at the time of enrollment
  The number of enrolled patients
Duration in minutes | Duration (minutes) will be measured each session up to 12 weeks.
  The investigators will determine if the delivery of a virtual physical activity program is feasible by tracking the number of minutes spent in the warm up, activity and cool-down.
Heart Rate | Intensity ( heart rate) will be measured each session up to 12 weeks.
  In order to objectively measure the intensity level and volume of PA during the activity sessions, participants will wear accelerometers on their waist and a wrist-based heart rate will be used to intensity of PA in real-time.
Relative Rate of Perceived Exertion | Intensity (RPE) will be measured each session up to 12 weeks.
  Rate of perceived exertion (RPE) will be obtained from participants as a subjective measure of intensity.
Acceptability of the program by patients | Focus groups will be conducted up to 12 weeks.
  The virtual activities also need to enjoyable, so with the use of focus groups, patient acceptability of the program will be determined. Predetermined questions and prompts will be used, such as, "Describe a lesson or lessons you liked best. What are some lessons that were less enjoyable? What was the most difficult aspect of participating in PePA? In general, did the exercises feel like they provided the right amount of exertion, too intense, not intense enough? Was the duration of each session too long, too short or about right?". The focus group recording will be transcribed and themes will be identified in this qualitative analysis.
Adherence | Attendance will be measured each week up to 12 weeks. If the participant continues for a second round, adherence will be measured each week during the second intervention up to 12 weeks.
  The number of completing patients. This will be measured by counting the number of participants who completed the majority of the program for each round (i.e., 20 out of 24 sessions).

SECONDARY OUTCOMES:
Health-related quality of life (QL) | Change from baseline QL at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program with the following measure:
  Quality of life with the Pediatric Quality of Life Inventory General Well-Being Scale (PedsQL Inventory, 23 items). Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 3=25, 4=0. Higher scores reflect better outcomes.
Physical Activity Intention | Change from baseline physical activity intention at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Physical Activity (PA) intention with the PA Intention Inventory (6 items). The first 3 items ask about the number of days over the past week the participant engaged in PA for 60 minutes, the number of days PA was engaged which resulted in elevated heart rate, and the number of days that the participant engaged in resistance exercises. Responses range from 0-7 days with greater days indicating more activity.
  The last 3 questions ask the participant about his/her intention to engage in PA outside of school, participate in PA which makes him/her breathe hard in the next 2 weeks and if s/he expects to exercise outside of school that makes him/her breathe hard in the next 2 weeks. Answers correspond to 0=strongly agree, 1=agree, 2= not sure, 3=disagree, 4=strongly disagree. Scores range from 0-12, with lower scores reflecting better outcomes.
Social Support | Change from baseline Social Support at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Social support toward PA from friends and parents (Social Support Questionnaire, 8 items). Items are answered with very often (0), often (1), neutral (2), sometimes (3) or never (4). Scores range from 0 to 32. Lower scores represent better outcomes.
Fatigue | Change from baseline Fatigue at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Fatigue using the PedsQL Multidimensional Fatigue Scale Questionnaire (18 items). Items are transformed to a 0-100 scale, where 0=100, 1=75, 3=25, 4=0. Scores are averaged (divided by 18) and range from 0-100. Higher scores indicate fewer problems.
Depression | Change from baseline Depression at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Depression using the Children's Depression Inventory (12 items). Items 1, 3-6, 8, 10-12 correspond to emotional problems. Items 2, 7, 9, 13-17 correspond to function problems. Reverse scoring is used for items 2, 7, 13, 14, 16. Higher scores indicate greater problems. Scores are compared to normative ranges (0-39+), which are age- and sex-dependent.
Cardiorespiratory endurance | Change from baseline Cardiorespiratory Endurance at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Cardiorespiratory endurance using the 6-minute walk test (ml/kg/min).
Flexibility | Change from baseline Flexibility at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Range of motion using goniometry (degrees).
Hand Strength | Change from baseline Hand Strength at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Hand strength will be measured with hand-held dynamometry (kg).
Muscular Strength | Change from baseline Muscular Strength at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  A manual muscle testing (scale that rates trace, poor, fair, good, normal performance) will be used to measure Muscular Strength.
Balance | Change from baseline Balance at 12 weeks.
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Balance using the Berg Balance Scale (14 items). Scores range from 0 to 56 with higher scores reflecting better outcomes.
Activity of daily living (ADL) | Change from baseline ADL at 12 weeks..
  The investigators will explore the trends of a virtual physical activity program on the following measure:
  Assessment of the ability to perform activities of daily living (ADL, QuickDASH Inventory, 11 items). Items are scored as no difficulty (1), mild difficulty (2), moderate difficulty (3), severe difficult (4), to unable to achieve (5). At least 10 items need to be completed and is measured on a scale of 0-100 with a higher score indicating greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Paulette Yamada Tamashiro, PhD, Principal Investigator — University of Hawaii
Locations (3):
- United States (3):
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - University of Hawaii at Manoa, Honolulu, Hawaii
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii

IPD SHARING:
Plan to Share IPD: Undecided
Since the number of subjects that will is small (n=12), IPD may be easily tracked to the patient themselves. If it is possible to mask / de-identify data, IPD may be shared at the conclusion of this study.

REFERENCES:
- [Background] Ouyang N, Cai R, Zhou X, Huang H, Qiu X, Liu K. Effects of a group-based physical activity program for pediatric patients with cancer on physical activity and symptom experience: A quasi-experimental study. Pediatr Blood Cancer. 2019 Nov;66(11):e27965. doi: 10.1002/pbc.27965. Epub 2019 Aug 12. PMID 31407493
- [Background] Honas JJ, Washburn RA, Smith BK, Greene JL, Cook-Wiens G, Donnelly JE. The System for Observing Fitness Instruction Time (SOFIT) as a measure of energy expenditure during classroom-based physical activity. Pediatr Exerc Sci. 2008 Nov;20(4):439-45. doi: 10.1123/pes.20.4.439. PMID 19168920
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Panepinto JA, Torres S, Bendo CB, McCavit TL, Dinu B, Sherman-Bien S, Bemrich-Stolz C, Varni JW. PedsQL Multidimensional Fatigue Scale in sickle cell disease: feasibility, reliability, and validity. Pediatr Blood Cancer. 2014 Jan;61(1):171-7. doi: 10.1002/pbc.24776. Epub 2013 Sep 13. PMID 24038960
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Quatman-Yates CC, Gupta R, Paterno MV, Schmitt LC, Quatman CE, Ittenbach RF. Internal consistency and validity of the QuickDASH instrument for upper extremity injuries in older children. J Pediatr Orthop. 2013 Dec;33(8):838-42. doi: 10.1097/BPO.0b013e3182a00688. PMID 23863415
- [Background] Rider BC, Conger SA, Ditzenberger GL, Besteman SS, Bouret CM, Coughlin AM. Examining the Accuracy of the Polar A360 Monitor. J Strength Cond Res. 2021 Aug 1;35(8):2165-2169. doi: 10.1519/JSC.0000000000003136. PMID 34398076
- [Result] Yamada PM, Centeio EC, Bantum EO, Cao S, Lopez GM. Informing the delivery of physical activity leadership for pediatric patients undergoing cancer treatment. International Journal of Kinesiology in Higher Education, Sept 2023. DOI: 10.1080/24711616.2023.2237427